CLINICAL TRIAL: NCT03425760
Title: A Cross-sectional Study of COPD and Symptom Variability in MEA Countries
Acronym: COPVAR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00105
Record Dates: First submitted 2018-01-22; First posted 2018-02-08 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional study aims at assessing stable GOLD C and D COPD patient's perception of daily and weekly symptoms variability and their impact on daily activities.

It will also explore the current practice in management of stable GOLD C and D COPD patients.

DETAILED DESCRIPTION:
1. Primary objective: To assess perception of daily and weekly variability of symptoms in stable GOLD C and D COPD patients and their impact on daily life activities
2. Secondary objectives:

   * To describe the current treatment practice for the management of GOLD C and D COPD in MEA countries and their adherence to the GOLD 2015 guidelines
   * To compare patients' perception of symptoms variability and their impact on activities between Gold categories C and D
   * To identify demographic, behavioral and clinical factors associated with symptoms variability.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion have to fulfill all of the following criteria:

  1. Stable GOLD C or D COPD patient under maintenance treatment, over 45 years, who provided signed informed consent;
  2. COPD diagnosis documented by spirometry performed in the past 12 months with an FEV1/FVC < 0.7 and an FEV1 < 50% predicted.

Exclusion Criteria:

Patients are not eligible for inclusion if they meet one of the following criteria:

1. Patient with an ongoing COPD exacerbation*;
2. Patient who has experienced an exacerbation* in the previous 3 months;
3. History of asthma, allergic rhinitis, lung cancer or any other significant respiratory disease, such as tuberculosis, lung fibrosis or sarcoidosis;
4. Inability to understand the study related questions;
5. Mentally disabled patient or unable to read and write;
6. Pregnant.
7. Current participation in a clinical trial;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stable GOLD C or D COPD patient under maintenance treatment, over 45 years
Sampling Method: Non-Probability Sample
Enrollment: 3254 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Perception of symptoms variability in Chronic obstructive pulmonary disease(COPD) patients | 1 Year
  Mean score of Morning Activities and Symptoms Questionnaires (MASQ). MASQ is a patient-reported outcome instrument developed to measure morning activities and morning symptoms. The MASQ consist of two parts that captures instant symptoms through the Global Chest Symptoms Questionnaire (GCSQ), and morning activities through the Capacity of Daily Living during the morning (CDLM) questionnaire. Each item is rated on a 5 point Likert scale, from 0 (not at all) to 4 (extremely), the total score being calculated as the average score of the two questions. Score Range a score ranging from 0 (so difficult that the activity could not be carried out by the patient on their own) to 5 (activity was not at all difficult to carry out).
Impact of symptom variability on daily life activities of Chronic obstructive pulmonary disease(COPD) Patients | 1 Year
  Percentage of patients whose daily activities are affected as captured in the Chronic obstructive pulmonary disease(COPD) Assessment Test(CAT). CAT IS a questionnaire that assesses the impact of COPD (cough, sputum, dyspnoea, chest tightens) on health status. There are eight questions with a scale of 1 to 5. Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life. The difference between stable and exacerbation patients was five units. No target score represents the best achievable outcome.

SECONDARY OUTCOMES:
Current treatment practice for the management of COPD in Middle East Africa countries and their adherence to The Global Initiative for Chronic Obstructive Lung Disease(GOLD 2015) guidelines | 1 Year
  Patients whose treatment is adherent with The Global Initiative for Chronic Obstructive Lung Disease(GOLD) 2015 in Percentage

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=24814&filename=Synopsis_COPVAR_CSR_AZ_version_1.2_20-June-2018.pdf